CLINICAL TRIAL: NCT01732848
Title: A Follow-up Evaluation for Safety in Subjects Who Participated in a Phase 1 Study With BMS-986094 (INX-08189)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI472-013
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Healthy; Hepatitis C
Keywords: Volunteers
MeSH Terms: conditions — Hepatitis C | interventions — BMS-986094

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects treated with BMS-986094/INX-08189: Subjects who participated in a clinical trial in which at least 1 dose of BMS-986094/INX-08189 was administered
  Interventions: Drug: BMS-986094/INX-08189
- Subjects treated with Placebo matching BMS-986094/INX-08189: Subjects who participated in a clinical trial in which at least 1 dose of Placebo matching BMS-986094/INX-08189 was administered
  Interventions: Drug: Placebo matching BMS-986094/INX-08189

INTERVENTIONS:
Drug: BMS-986094/INX-08189
  Other Names: Observational study - No Intervention subjects were previously treated with BMS-986094/INX-08189
  Groups: Subjects treated with BMS-986094/INX-08189
Drug: Placebo matching BMS-986094/INX-08189
  Other Names: Observational study - No Intervention subjects were previously treated with Placebo matching BMS-986094/INX-08189
  Groups: Subjects treated with Placebo matching BMS-986094/INX-08189

SUMMARY:
The purpose of this study is to determine the rate of kidney or heart impairment, if any, in subjects who received BMS-986094 (INX-08189) in Phase 1 clinical trials

ELIGIBILITY:
Inclusion Criteria:

* Healthy and hepatitis C virus (HCV)-infected subjects who participated in prior Phase 1 trial with BMS-986094/INX-08189 and:

  1. Received at least 1 dose of INX-08189 or
  2. Received placebo in studies for HCV-infected subjects (INH-189-002 or INH-189-006)
* Age 18 or older

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who participated in prior trial with BMS-986094/INX-08189 and received at least 1 dose of INX-08189 or placebo in trials INH-189-002 or INH-189-006
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Rate of renal impairment among subjects exposed to BMS-986094 in the Phase 1 program that meet the predefined criteria for impaired renal function and require referral to a nephrologist | Up to Day 90
Rate of cardiac impairment among subjects exposed to BMS-986094 in the Phase 1 program that meet the predefined criteria for impaired cardiac function and require referral to a cardiologist | Up to Day 90

SECONDARY OUTCOMES:
Changes in the electrocardiographic parameters observed in association with prior exposure to single and multiple oral doses of BMS-986094 compared to pre-exposure electrocardiograms (ECGs) | Baseline (pre-dose Day 1 ECG from parent study) and By Day 30
Abnormalities in cardiac ejection fraction (EF) as determined by trans-thoracic echocardiogram that may be associated with prior exposure to single or multiple oral doses of BMS-986094 | By Day 90
Abnormalities in B-type-natriuretic peptide (BNP) levels that may be associated with prior exposure to single or multiple oral doses of BMS-986094 | By Day 30
Changes in serum creatinine levels compared to pre-exposure levels that may be associated with prior exposure to single or multiple oral doses of BMS-986094 | Baseline (Day 1 from parent study) and By Day 14
Abnormalities in urinary albumin excretion that may be associated with prior exposure to single or multiple oral doses of BMS-986094 | By Day 7
Presence of signs, symptoms or medical history suggestive of heart failure or renal failure that may have been observed since last exposure to BMS-986094 | By Day 90
Abnormalities in creatine phosphokinase (CPK) and creatine phosphokinase-metabolic (CPK-MB) levels that may be associated with prior exposure to single or multiple doses of BMS-986094 | By Day 30
Abnormalities in troponin levels that may be associated with prior exposure to single or multiple doses of BMS-986094 | By Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (4):
  - Local Institution, Los Angeles, California
  - Prism Research, Saint Paul, Minnesota
  - New Orleans Center For Clinical Research - Knoxville, Knoxville, Tennessee
  - Local Institution, San Antonio, Texas
- Local Institution, San Juan, Puerto Rico

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx